CLINICAL TRIAL: NCT07024836
Title: PRecision biomArker-Guided MAnagement of TuberculosIs Contacts: a Discrete Choice Experiment
Acronym: PRAGMATIC-DCE
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 175542
Record Dates: First submitted 2025-05-16; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis (TB)
Keywords: preference; discrete choice experiment; qualitative; latent tuberculosis infection
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient participants for qualitative stage (stage 1): Semi-structured interviews will first be conducted among 20-30 people undergoing testing for latent tuberculosis infection, as part of routine clinical screening programmes (Stage 1).
- Patient participants for discrete choice experiment (stage 2): 200 patients will then undertake a quantitative discrete choice experiment to evaluate preferences and trade-offs that influence acceptance of preventive TB treatment.
- Healthcare worker participants for discrete choice experiment (stage 2): 200 healthcare workers will also undertake a quantitative discrete choice experiment to evaluate preferences and trade-offs that influence recommendation of preventive TB treatment.

SUMMARY:
This study is part of a broader programme of work to develop and pilot a randomised-controlled trial of new tests to identify people who will benefit most from preventive treatment for tuberculosis (TB). The aim of the current study is to explore factors affecting patient decisions to start preventive treatment. The specific objectives are to understand how patients make decisions about preventive treatment initiation for TB (stage 1); and to design and conduct a "discrete choice experiment" survey to further evaluate preferences (stage 2).

DETAILED DESCRIPTION:
We will perform up to 30 semi-structured interviews among people undergoing testing for latent TB infection, as part of routine clinical screening programmes (stage 1). Adults (aged ≥18 years) who have been or are being tested for LTBI in routine clinical services will be eligible for inclusion through purposive sampling. The findings from the qualitative study will then be used to inform the a discrete choice experiment (DCE). The DCE will be conducted to quantify the trade-off between future TB risk and preventive treatment acceptance, from patient and healthcare provided perspectives (stage 2).

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged ≥18 years) who have been tested for latent TB infection in routine clinical services, or are eligible for testing. Eligible people for testing include migrants from countries with high TB incidence (entered UK within 5 years), people with recent contact with a person with TB disease, and people eligible for LTBI screening prior to starting immunosuppression or through occupational health testing.

Exclusion Criteria:

* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Adults tested, or eligible for testing, for latent tuberculosis infection in routine clinical services.
  2. Nurses, doctors or allied health professionals who have any experience of testing or treatment for TB or latent TB infection in UK services.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Preventive treatment acceptance | Baseline
  Discrete choice experiment data will be analysed to evaluate the primary outcome of preventive TB treatment acceptance in the survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Whittington Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data from the discrete choice experiment will be made publicly available at the time of peer-reviewed publication.
Time Frame: Indefinitely from the time of peer-reviewed publication.
Access Criteria: The anonymised discrete choice experiment data will be publicly available